CLINICAL TRIAL: NCT04212988
Title: Effect of Cerebral Oxygen Saturation Interventionon Postoperative Delirium After Cardiac Surgery
Brief Title: Effect of Cerebral Oxygen Saturation Intervention
Acronym: ECOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJTU1AF-CRF-2017-009
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: single blind
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the trial group (Experimental): The interwention process will be started once the SCO2 value below ideal levels (80% of the basic level or 50% of absolute value), by adjusting the position of extracorporeal circulation arteriovenous catheter, balancing arterial pressure, increasing oxygen supply , adjusting pump speed ,etc.
  Interventions: Procedure: Increase the SCO2 value
- the control group (Placebo Comparator): In control group patients, only place the probe for NIRS monitor.
  Interventions: Procedure: Increase the SCO2 value

INTERVENTIONS:
Procedure: Increase the SCO2 value — The interwention process will be started once the SCO2 value below ideal levels (80% of the basic level or 50% of absolute value), by adjusting the position of extracorporeal circulation arteriovenous catheter, balancing arterial pressure, increasing oxygen supply , adjusting pump speed ,etc.

SUMMARY:
Postoperative delirium (POD) is a common complication after cardiac surgery,and the pathogenesis is considered imbalance of cerebral oxygen. It may induce the POD incidence by monitering and intervening the low cerebral oxygen desaturation(SCO2) in cardiac surgery .Near infrared spectroscopy (NIRS) will be used for monitering the cerebral oxygen levels.140 case will be included and divided in to trial and control group. The primary outcome is POD In 72 hours after the surgery , which is assessed according to delirium scale .

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a common complication after cardiac surgery. Imbalance of cerebral oxygen supply and demand is one of the pathogenesis of postoperative delirium. The perioperative cerebral oxygen levels and postoperative delirium highly correlated, while as a high incidence of cerebral oxygen desaturation(SCO2) in cardiac surgery, especially in extracorporeal circulation. Near infrared spectroscopy (NIRS) can monitor the SCO2 continuously, noninvasively, simultaneously on bilateral cerebral hemisphere, and monitoring will not restricted by extracorporeal circulation.Using NIRS to moniter and intervene thecerebral oxygen levels in extracorporeal circulation of heart surgery patients ,thereby reducing the incidence of postoperative delirium. This hypothesis has a very important clinical value.

This study intends to include 140 patients, who requires extracorporeal circulation cardiac surgical treatment. All cases will be divided into trial group and control group preoperative follow-up.Two groups of patients in surgery will be both performed the investigator's existing standerd monitoring and surgery process.

The trial group cases will be given NIRS monitoring in the whole surgical procedure. And once the SCO2 value below ideal levels (80% of the basic level or 50% of the absolute value), the intervention process will be started immediately to correct the low cerebral oxygen status, by adjusting the position of extracorporeal circulation arteriovenous catheter, stabilizing the mean arterial pressure, increasing oxygen supply and , adjusting the pump speed, etc. The control group cases will be only placed the probe of NIRS moniter.

In 72 hours after the surgery , all patients will be assessed POD by cardiac surgery intensivecare unit(CICU) physicians according to delirium scale .

This project intends to research monitoring brain oxygen supply and intervention can reduce the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Participate and sign the informed consent voluntary;
2. Over 18 years of age;
3. Who recieve the heart surgery under extracorporeal circulation;
4. Able to communicate and abey the experimental requirements well .

Exclusion Criteria:

1. Refused to sign a consent form;
2. Less than 18 years of age;
3. With history of nervous, mental, and cerebrovascular disease;
4. With history of alcohol or apsychiatric drug addiction;
5. Can't cooperate the evaluation: dementia, dysaudia, visually impaired , etc;
6. Critically diseases: severe liver and kidney dysfunction, cardiac shock or IABP placement status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
the incidence of POD | 3 days after sugery
  the incidence of postoperative delirium in the cases after 3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- FirstXianJiaotongU, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No